CLINICAL TRIAL: NCT05277246
Title: Effect of Using Different Concentrations of NaOCI on IL-8 Level During Endodontic Treatment of Teeth With Irreversible Pulpitis
Brief Title: Effect of Using Different Concentrations of NaOCI on IL-8 Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Esin Özlek, Asis.Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/15.12.2021
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Irreversible Pulpitis
Keywords: Gingival cervicular fluidi; IL-8

STUDY DESIGN:
Intervention Model Description: Group 1; 2 ml of 1% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Group 2: 2 ml of 2.5% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Group 3; 2 ml of 5.25% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1% NaOCIL (Active Comparator): 2 ml of 1% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Interventions: Other: Irrigant concentration; Drug: NaOCI
- 2.5% NaOCI (Active Comparator): 2 ml of 2.5% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Interventions: Other: Irrigant concentration; Drug: NaOCI
- 5.25% NaOCI (Active Comparator): 2 ml of 5.25% NaOCl solution will be used as irrigation solution at every file change during root canal preperation .2 ml dental injector and 27 gauge thickness dental needle tip will be used for irrigation . The tip of the cannula will be adjusted to reach two-thirds of the working length.
  Interventions: Other: Irrigant concentration; Drug: NaOCI

INTERVENTIONS:
Other: Irrigant concentration — The success of endodontic treatment is directly related to infection control. In successful endodontic treatment, it is necessary to perform an ideal irrigation both in order to gain a better understanding of the complex anatomical structure of the root canals and to increase the efficiency of the instruments and methods used during the canal preparation. Sodium hypochlorite (NaOCl) solution is the standard irrigation agent for cleaning and disinfection of root canal. In this study, the effect of NaOCI on level of IL-8 different concentration will be evaluated.
Drug: NaOCI — NaOCI

SUMMARY:
The objective is to compare various concentrations of NAOCL during Root canal treatment and their effect on IL-8 at the gingival crevicular fluid. Despite the current advancement of beneficial endodontic diagnostic methods, such as pulp sensitivity tests and periapical radiographs, clinical outcomes do not always correspond with the arrangement of the histological condition of the pulp. At this point, the need for other ways to help diagnose pathological pulpal disease has arisen. This situation has influenced researchers to use molecular evaluation as an alternative route in endodontic diagnosis. Biomarkers, functional at the cellular and molecular level, are crucial elements within the pathological process. Detection of molecular markers is considered an ancillary method for diagnosing the pathological condition of the pulp tissue.An increase in inflammatory cells in the carious or traumatized dentinal pulp complex has been reported. In the presence of bacteria, immune cells produce interleukin-6 (IL6), interleukin-8 (CXCL8), and tumor necrosis factor-alpha (TNF) in the pulp. Interleukin-8 is frequently expressed in endothelial cells of inflamed pulp and rarely in the normal pulp. Karapanou et al. (2008) revealed that interleukin-8 was more greatly released in teeth with irreversible pulpitis than in the control group in a research in which gingival crevicular fluid with acute pulpitis was analyzed. the pulp tissue and gingival crevicular fluid of teeth with symptomatic irreversible pulpitis were dramatically augmented by these indicators compared with healthy teeth. Furthermore, they concluded that the levels of NKA, SP, IL8, and MMP8 in the gingival crevicular fluid decreased one week after endodontic treatment of teeth with pulpitis. Subsequently, it has been reported that patients with symptomatic irreversible pulpitis with high initial pain scores have higher levels of SP, IL8, and MMP8 in the pulp tissue samples than those with low pain scores.It is recommended to use NaOCl concentration between 0.5% and 5.25% as an irrigation solution in root canal treatment (6). The effectiveness of NaOCl increases with increasing concentration, but its toxicity is known to be proportional to concentration.

Therefore, there is no consensus on the optimal concentration of NaOCL. When articles were reviewed, it was found that inflammation of the pulp and biomarker levels are correlated. For this reason, we believe that whether or not NaOCl solution at various concentrations causes inflammation can be analyzed by the level of IL-8. Upon review of the literature, it was found that no studies investigated the influence of NaOCl solution on biomarkers in the gingival crevicular fluid. The research described below contributes to the literature on the optimal concentration of NaOCl to use.

DETAILED DESCRIPTION:
The study is to be carried out in 84 medically fit patients, aged 18-50 years, who were diagnosed and followed up at Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Endodontics, (The number of patients was determined according to "power analysis.") Lower first and second molars (36,37,46,47) diagnosed with irreversible pulpitis will be included in the study as an experimental group.

As the control group, the contralateral teeth of the related teeth will be evaluated. Patients with periapical lesions and open apex teeth will not be included in the study group. Before treatment, patients will be asked to determine their pain level according to a 0-10 VAS scale, and this value will be recorded for comparison with post-treatment. Teeth (experimental and control ) to be sampled from the gingival crevicular fluid will be isolated with a cotton roll and saliva ejector.

The supragingival plaque will be carefully removed using a curette. The teeth to be inspected will be dried with air for 10 seconds. A Periopaper strip (Oraflow, Smithtown, NY, USA) will be placed in the interproximal mesial gingival sulcus of the affected tooth until slight resistance is confronted and is removed after 1 min. Samples contaminated with blood or saliva will not be involved in the study. All collected periopaper strips will be placed in 1.5 ml Eppendorf tubes (Labosel, Istanbul, Turkey) and stored at -80 ° C until analysis.

After applying 2ml local anesthesia (Maxicaine DS strong (Vem, İstanbul, Türkiye)), the access cavity will be opened with diamond bur. The working length will be determined using the apex locator (DentsplyMaillefer, UK) and the radiographic x-ray by placing a K file #15 (Mani Inc, Tochigi, Japan) into the root canals until the apical constriction.

The shaping process of the root canals will be accomplished by ProTaperNext (DentsplyMaillefer, Baillagues, Switzerland) up to the X3 instrument as standard in each patient. The study will be randomly divided into 3 groups (n= ) according to the irrigation solution used during shaping (G1: 1% NaOCl; G2: 2.5% NaOCl; G3: 5.25% NaOCl). 2 ml of irrigation solution will be applied after each file.

A 2 ml dental injector with a 27 gauge dental needle will be used; the tip of the needle will be adjusted to reach two-thirds of the working length. For the final irrigation of the root canals that have completed the shaping process, 5 ml of 17% EDTA solution and NaOCl solution will be used, respectively. Later on, the canals will be dried with sterile paper points.

Root canals will be obturated with sterile gutta-perchas and AH+ (Dentsply De Trey, Konstanz, Germany) root canal sealer using the single cone technique.

Finally, the teeth will be restored using composite. One week after treatment, the patient will be called for a follow-up appointment.

The patients will be asked to determine the pain level according to the VAS scale, and it will be recorded. A specimen of gingival crevicular fluid will be taken from the root canal treated teeth in the same manner as at the commencement and stored. The amount of IL-8 in the gingival crevicular fluid will be measured with an enzyme-linked immunoassay (ELISA) kit (Cayman, Ann Arbor, MI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons between the ages of 18 and 45 years
* Mandibular molar teeth that were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Patients who are taken analgesic inflammatory drugs with in the last 12 hours
* Pregnancy or lactation
* Teeth with periodontal diseases
* Teeth with sensitive to percussion and palpation
* Teeth with root resorption
* Teeth with immature/open apex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
IL-8 Level | 6 months
  Concentration of IL-8 in GCF

IPD SHARING:
Plan to Share IPD: No